CLINICAL TRIAL: NCT04736381
Title: Impact of the Microbiota on the Likelihood of Renal Graft Rejection
Acronym: MERRLIN
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C 19-53
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Rejection
Keywords: Microbiota; Belatacept; Second signal inhibitor
MeSH Terms: interventions — Abatacept; Basiliximab; Mycophenolic Acid; Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Kidney transplanted patients treated with Nulojix: Patients treated with Simulect as induction, and with Nulojix®, mycophenolic acid and steroids as maintenance therapy during the first year of kidney transplant.
  Interventions: Drug: Belatacept Injection [Nulojix]

INTERVENTIONS:
Drug: Belatacept Injection [Nulojix] — Drugs administrated are part of the usual care
  Other Names: Simulect; Mycophenolate mofetil; Steroid

SUMMARY:
Identification of a bacterial signature in the blood or stool that may be associated with acute rejection in patients treated with Nulojix during their first year of transplant.

DETAILED DESCRIPTION:
Gut microbiota as well as the signature of the 16S plasma bacterial DNA and bacterial metabolites of patients on the date of transplantation and during the first year after transplantation will be analyzed. The phenotype of the patients' T lymphocytes will be analyzed at the same time. These data will be correlated with the occurrence of acute cell rejection during the first year of transplantation

ELIGIBILITY:
Inclusion Criteria:

* Patients called for a kidney transplant
* Induction therapy with Simulect, maintenance therapy with Nulojix, mycophenolate acid and steroids
* Patient having signed the informed consent

Exclusion Criteria:

* Multiple grafts combined or sequential
* Induction therapy with polyclonal antibodies
* HIV or active viral infection such as hepatitis B or C
* Active bacterial infection
* Pregnancy or breastfeeding at time of inclusion
* Patient unable to express their consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients treated with Simulect as induction, and with Nulojix®, mycophenolic acid and steroids as maintenance therapy during the first year of kidney transplant.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Acute rejection occurence | 1 year or rejection
  Occurence of cellular rejection according to the BANFF 2017

SECONDARY OUTCOMES:
Gut and circulating microbiota | 1 year or rejection
  16S DNA sequencing
Lymphocyte phenotype | 1 year or rejection
  CD3+CD4+CD57+PD1-, CD3+CD8+CD28low, CD3+CD8+CD45RA phenotype
Glomerular filtration rate | 1 year or rejection
  CDK-EPI creatinine equation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Durrbach, MD-PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (9):
- France (9):
  - Nephrologie transplantation CHRU Besançon, Besançon
  - Néphrologie, hémodialyse, aphérèses, transplantation rénale, La Tronche
  - Nephrologie transplantation CHRU Nantes, Nantes
  - Nephrologie transplantation CHU Saint Louis Paris, Paris
  - Nephrologie transplantation CHU Pitié Salpetriere Paris, Paris
  - Nephrologie hôpital Henri-Mondor, Paris
  - Nephrologie transplantation CHRU Poitiers, Poitiers
  - Nephrologie transplantation CHRU Toulouse, Toulouse
  - Nephrologie transplantation CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincenti F, Blancho G, Durrbach A, Friend P, Grinyo J, Halloran PF, Klempnauer J, Lang P, Larsen CP, Muhlbacher F, Nashan B, Soulillou JP, Vanrenterghem Y, Wekerle T, Agarwal M, Gujrathi S, Shen J, Shi R, Townsend R, Charpentier B. Five-year safety and efficacy of belatacept in renal transplantation. J Am Soc Nephrol. 2010 Sep;21(9):1587-96. doi: 10.1681/ASN.2009111109. Epub 2010 Jul 15. PMID 20634298
- [Background] Durrbach A, Pestana JM, Pearson T, Vincenti F, Garcia VD, Campistol J, Rial Mdel C, Florman S, Block A, Di Russo G, Xing J, Garg P, Grinyo J. A phase III study of belatacept versus cyclosporine in kidney transplants from extended criteria donors (BENEFIT-EXT study). Am J Transplant. 2010 Mar;10(3):547-57. doi: 10.1111/j.1600-6143.2010.03016.x. PMID 20415898